CLINICAL TRIAL: NCT00331994
Title: Efficacy Evaluation of Enterogermina, 2 Billion Bacillus Clausii Spores, on Eradication of Small Intestinal Bacterial Overgrowth: a Randomised, Parallel-group, Open Study.
Brief Title: EFESO - EFficacy Enterogermina Small Intestinal Bacterial Overgrowth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Medical Director, Sanofi-aventis aministrative office
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0161; EudraCT # : 2005-004934-42
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — clausin peptide, Bacillus clausii; Metronidazole

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Bacillus clausii
- 2 (Active Comparator)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Bacillus clausii — 3 bacillus clausii vials/day for one month
  Arms: 1
Drug: Metronidazole — 3 Metronidazole tablets/day for one week
  Arms: 2

SUMMARY:
Primary objective: to assess the efficacy of Bacillus clausii versus metronidazole in the eradication of the small intestinal bacterial overgrowth, 30 days after the end of treatment.

Secondary objective: to assess the efficacy of Bacillus clausii versus metronidazole in avoiding recurrence of the small intestinal bacterial overgrowth, 90 days after the end of the treatment; to assess the efficacy of Bacillus clausiiversus metronidazole in improving irritable bowel syndrome -related symptoms; to assess the efficacy of Bacillus clausii versus metronidazole in the satisfactory relief of overall irritable bowel syndrome symptoms and of abdominal discomfort or pain; to assess the efficacy of Bacillus clausii versus metronidazole in improving irritable bowel syndrome quality of life.

ELIGIBILITY:
Inclusion criteria:

* Irritable bowel syndrome patients with small intestinal bacterial overgrowth (based on positive lactulose or glucose hydrogen breath test)
* Patients able to maintain their usual diet and lifestyle during the course of the study.

Exclusion criteria:

* Pregnancy or breast-feeding
* Major concomitant diseases (including tumours and hepatic and/or renal insufficiency)
* Inflammatory bowel diseases
* History of intestinal surgery (except cholecystectomy and appendectomy)
* Use of antibiotic, laxative, antidiarrheic drugs or probiotics (medications or dietetic supplements) in the last month prior to study entry
* Hypersensibility to the investigational product and reference drug
* Clinical evidence of relevant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurologic or of any disease that may interfere with the patient successfully completing the trial or the objectives of the trial
* Eating disorders such as anorexia or bulimia, and/or psychosis, schizophrenia, mania or major psychiatric illness needing pharmacological treatment. Well-compensated depression does not exclude a potential patient
* Participation to a trial in the previous three months
* Drug or alcohol abuse
* Subjects with unstable personality or not able to be compliant with the study procedures

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
eradication rate of the small intestinal bacterial overgrowth | 30 days after the end of the treatment.

SECONDARY OUTCOMES:
avoiding recurrence of the small intestinal bacterial overgrowth | 90 days after the end of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Milan, Italy